CLINICAL TRIAL: NCT07049445
Title: A Randomized Controlled Trial on the Effect of Music Activities on Depression and Sleep Quality in Frail Older Adults
Brief Title: Effect of Music Activities on Depression and Sleep Quality in Frail Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Chung Hsing University (Other)
Responsible Party: Principal Investigator, Chia-Te Chen, Assistant Professor, National Chung Hsing University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-ER-114-152
Record Dates: First submitted 2025-06-22; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Depression; Sleep Quality; Frailty
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders; Frailty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Behavioral: Music Activity Program
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Music Activity Program — Participants in the experimental group will receive the standard day care center activities plus a music activity intervention. The music activity consists of pre-recorded video sessions conducted twice a week, each lasting one hour, for a total duration of 8 weeks.
  Arms: Experimental Group

SUMMARY:
This study aims to examine the effects of music activities on depression and sleep quality among frail older adults, and to develop a standardized music activity protocol suitable for use in adult day care centers. A randomized controlled trial (RCT) design will be used. Participants will be recruited from 4 to 5 adult day care centers and randomly assigned to either an intervention group (receiving music activities twice per week, one hour per session, for eight weeks) or a control group (receiving only routine activities). Depression and sleep quality will be measured at baseline, week 4, and week 8. Assessments will include validated questionnaires and the index of osteoporotic fractures. Data analysis will evaluate the effectiveness of music activities in improving depression and enhancing sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Aged 60 years or older.
  2. Currently receiving services at an adult day care center.
  3. Frailty score ≥1 based on the Study of Osteoporotic Fractures (SOF) index.
  4. Geriatric Depression Scale (GDS-15) score ≥5 or Pittsburgh Sleep Quality Index (PSQI) score ≥5.
  5. Clear consciousness and able to communicate in Mandarin or Taiwanese.

Exclusion Criteria:

1. Severe hearing or visual impairments.
2. Diagnosed with severe psychiatric disorders or dementia.
3. Unable to participate in group activities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Geriatric Depression Scale-15 (GDS-15) | At baseline, week 4, and week 8
  The Geriatric Depression Scale-15 (GDS-15) is a self-report questionnaire used to assess depressive symptoms in older adults. It consists of 15 yes/no questions. Total scores range from 0 to 15, with higher scores indicating more severe depressive symptoms. A score of ≥5 is suggestive of depression. The scale is widely used and validated for older populations.
Pittsburgh Sleep Quality Index (PSQI) | At baseline, week 4, and week 8
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month interval. It includes 19 items generating 7 component scores (e.g., sleep latency, sleep duration), which are summed to yield a global score ranging from 0 to 21. Higher scores indicate poorer sleep quality. A global score >5 suggests significant sleep disturbances.

CONTACTS AND LOCATIONS:
Locations (1):
- huajiale Day Care Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data due to privacy considerations.

REFERENCES:
- [Background] Chu H, Yang CY, Lin Y, Ou KL, Lee TY, O'Brien AP, Chou KR. The impact of group music therapy on depression and cognition in elderly persons with dementia: a randomized controlled study. Biol Res Nurs. 2014 Apr;16(2):209-17. doi: 10.1177/1099800413485410. Epub 2013 May 2. PMID 23639952
- [Background] Chen CY, Wu SC, Chen LJ, Lue BH. The prevalence of subjective frailty and factors associated with frailty in Taiwan. Arch Gerontol Geriatr. 2010 Feb;50 Suppl 1:S43-7. doi: 10.1016/S0167-4943(10)70012-1. PMID 20171456
- [Background] Chen CT, Tung HH, Fang CJ, Wang JL, Ko NY, Chang YJ, Chen YC. Effect of music therapy on improving sleep quality in older adults: A systematic review and meta-analysis. J Am Geriatr Soc. 2021 Jul;69(7):1925-1932. doi: 10.1111/jgs.17149. Epub 2021 Apr 20. PMID 33880759
- [Background] Chen CT, Tung HH, Chen YC, Lee HF, Wang CJ, Lin WH. Depressive symptoms and nutritional status in the frail older adults. Arch Gerontol Geriatr. 2019 Jul-Aug;83:96-100. doi: 10.1016/j.archger.2019.03.023. Epub 2019 Mar 30. PMID 30991156
- [Background] Chen CT, Tung HH, Chen CW, Yang YR, Wang JL, Chang CM, Chen YC, Liang SH, Fan CH. Preventing functional decline in hospitalized older adults in medical ward: a best practice implementation project. JBI Evid Implement. 2024 Aug 1;22(3):271-280. doi: 10.1097/XEB.0000000000000411. PMID 38470609
- [Background] Chan MF, Chan EA, Mok E. Effects of music on depression and sleep quality in elderly people: A randomised controlled trial. Complement Ther Med. 2010 Jun-Aug;18(3-4):150-9. doi: 10.1016/j.ctim.2010.02.004. PMID 20688261
- [Background] Cervellin G, Lippi G. From music-beat to heart-beat: a journey in the complex interactions between music, brain and heart. Eur J Intern Med. 2011 Aug;22(4):371-4. doi: 10.1016/j.ejim.2011.02.019. Epub 2011 Mar 22. PMID 21767754
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Bilotta C, Nicolini P, Case A, Pina G, Rossi S, Vergani C. Frailty syndrome diagnosed according to the Study of Osteoporotic Fractures (SOF) criteria and adverse health outcomes among community-dwelling older outpatients in Italy. A one-year prospective cohort study. Arch Gerontol Geriatr. 2012 Mar-Apr;54(2):e23-8. doi: 10.1016/j.archger.2011.06.037. Epub 2011 Aug 25. PMID 21871675